CLINICAL TRIAL: NCT05296655
Title: Validity and Reliability of a Kazakh Version of Reflux Symptom Index
Brief Title: Kazakh Version of Reflux Symptom Index
Status: Completed | Type: Observational
Sponsor: Kazakh Medical University of Continuing Education (Other)
Collaborators: Asfendiyarov Kazakh National Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 14-2020/1
Record Dates: First submitted 2022-03-17; First posted 2022-03-25 (Actual); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Laryngopharyngeal Reflux Symptoms; Laryngopharyngitis Chronic; Gastro Esophageal Reflux Disease
Keywords: Laryngopharyngeal Reflux; Laryngopharyngeal Reflux Symptoms; Laryngitis; Laryngopharyngitis Chronic; Gastro Esophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux; Laryngopharyngeal Reflux; Laryngitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Laryngopharegeal reflux symptoms patients: patients with symptoms of laryngopharyngeal reflux detected at an outpatient appointment with an ENT doctor
  Interventions: Other: Reflux Symptom Index Inventory (diagnostic survey); Other: Reflux finding score
- Asymptomatic laryngopharegeal reflux patients: patients without symptoms of laryngopharyngeal reflux who applied for an appointment with an otorhinolaryngologist
  Interventions: Other: Reflux Symptom Index Inventory (diagnostic survey)

INTERVENTIONS:
Other: Reflux Symptom Index Inventory (diagnostic survey) — Kazakh versions of the Reflux Symptom Index Inventory will be filled patients
  Other Names: RSI
Other: Reflux finding score — laryngoscopy with a score RFS
  Other Names: RFS
  Groups: Laryngopharegeal reflux symptoms patients

SUMMARY:
Reflux symptoms index (RSI) were developed to identify a clinical index of suspicion for laryngopharyngeal reflux (LPR) in patients with ear, nose, and throat symptoms. RSI is an efficient diagnostic tool for LPR/ It is easy to use, even for those who know little about LPR. It does not require special equipment or examinations and is inexpensive. Thus, it can be considered highly efficient and cost-effective. The study will focus on translating and testing the RSI into Kazakh language and comparing its results in healthy people and people with laryngopharyngeal reflux.

ELIGIBILITY:
Inclusion Criteria:

* Patient's informed consent;
* Age: 18-74 years old;
* No serious somatic diseases;
* Patients with complaints of sore throat, coughing, burning sensation in the throat, coughing, frequent sore throat, difficulty swallowing, lump in the throat, foreign body feeling in the throat, voice changes, heartburn and belching;
* Diagnosis: Chronic pharyngitis;
* Chronic laryngitis.

Exclusion Criteria:

* Disagreement to participate in scientific research;
* Age: under 18 and over 74;
* Severe somatic diseases, organic lesions of the gastrointestinal tract and ENT organs;
* Patients with pulmonary pathologies;
* Patients with allergic manifestations (chronic or allergic rhinosinusitis and nasal polyposis);
* With diagnoses: Acute respiratory diseases;
* Patients with general neuralgic disorders;
* Pregnancy;
* Benign lesions of the vocal cords;
* Acid-suppressive therapy within 4 weeks prior to recruitment

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult female patients between 18 to 74 years of age with a laryngopharengeal symptoms and patients without symptoms of laryngopharyngeal reflux who applied for an appointment with an otorhinolaryngologist/
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2022-02-15 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
RSI Score at Baseline: | RSI Score at Baseline
  Patients will be asked to complete the Reflux Symptom Index questionnaire. An analysis of the results of the effectiveness of this method in patients with complaints of sore throat, coughing, burning sensation in the throat, cough, frequent sore throat, difficulty swallowing, lump in the throat, feeling of a foreign body in the throat, voice change, heartburn, belching will be carried out. The severity of the problem is calculated as the summation of all points. The problem is absent if the summation of points is 0. The problem is serious if the summation of points is 5. Total score ranges from 0-45; of which 0-12 is considered no laryngopharengeal reflux, above 13 points for the presence of laryngopharyngeal reflux.
RSI Score at Days 10-14 | Days 10-14
  Patients will be asked to complete the Reflux Symptom Index questionnaire. An analysis of the results of the effectiveness of this method in patients with complaints of sore throat, coughing, burning sensation in the throat, cough, frequent sore throat, difficulty swallowing, lump in the throat, feeling of a foreign body in the throat, voice change, heartburn, belching will be carried out. The severity of the problem is calculated as the summation of all points. The problem is absent if the summation of points is 0. The problem is serious if the summation of points is 5. Total score ranges from 0-45; of which 0-12 is considered no laryngopharengeal reflux, above 13 points for the presence of laryngopharyngeal reflux.
RFS Score at Baseline: | RFS Score at Baseline
  Device: Endoscopic laryngoscopy Video laryngoscopy and assessment of the presence / severity of the symptoms- Reflux finding score. Evaluation results range from 0 to 4, where 0 is an indicator of no problem, and 4 is an indicator of a serious problem. Total score ranges from 0-48; of which 0-6 is considered no laryngopharengeal reflux, above 7 points for the presence of laryngopharyngeal reflux.
RFS Score at Days 10-14 | Days 10-14
  Device: Endoscopic laryngoscopy Video laryngoscopy and assessment of the presence / severity of the symptoms - Reflux finding score and will be used as a gold standard of diagnosis of laryngopharengeal reflux. Evaluation results range from 0 to 4, where 0 is an indicator of no problem, and 4 is an indicator of a serious problem. Total score ranges from 0-48; of which 0-6 is considered no laryngopharengeal reflux, above 7 points for the presence of laryngopharyngeal reflux.
Reliability and validity of RSI at Baseline: | RSI Score at Baseline
  Reliability and validity of RSI at Baseline using Cronbach's alpha test to check the internal consistency for all the 9 items. Total score ranges from 0-45; of which 0-12 is considered no laryngopharengeal reflux, above 13 points for the presence of laryngopharyngeal reflux.
Reliability and validity of RSI at Days 10-14. | Days 10-14
  Reliability and validity of RSI at Days 10-14 using Cronbach's alpha test to check the internal consistency for all the 9 items. Total score ranges from 0-45; of which 0-12 is considered no laryngopharengeal reflux, above 13 points for the presence of laryngopharyngeal reflux.
Laryngopharyngeal reflux diagnosis at baseline | Baseline
  Video laryngoscopy and assessment of the presence / severity of the symptoms- Reflux finding score. Evaluation results range from 0 to 4, where 0 is an indicator of no problem, and 4 is an indicator of a serious problem. Total score ranges from 0-48; of which 0-6 is considered no laryngopharengeal reflux, above 7 points for the presence of laryngopharyngeal reflux.
Laryngopharyngeal reflux diagnosis at Days 10-14. | Days 10-14
  Video laryngoscopy and assessment of the presence / severity of the symptoms- Reflux finding score. Evaluation results range from 0 to 4, where 0 is an indicator of no problem, and 4 is an indicator of a serious problem. Total score ranges from 0-48; of which 0-6 is considered no laryngopharengeal reflux, above 7 points for the presence of laryngopharyngeal reflux.
Test - retest reliability of the RSI questtionaire | Days 10-14
  Test - retest reliability of the RSI questtionaire at Days 10-14. Test-retest reliability coefficients vary between 0 and 1, where:
  1 : perfect reliability,
  0.9: excellent reliability, 0.8 < 0.9: good reliability, 0.7 < 0.8: acceptable reliability, 0.6 < 0.7: questionable reliability, 0.5 < 0.6: poor reliability, < 0.5: unacceptable reliability, 0: no reliability. On this scale, a correlation of .9(90%) would indicate a very high correlation (good reliability) and a value of 10% a very low one (poor reliability).
Test - retest reliability of the RFS | Days 10-14
  Test - retest reliability of the RFS questtionaire at Days 10-14. Test-retest reliability coefficients vary between 0 and 1, where:
  1 : perfect reliability,
  0.9: excellent reliability, 0.8 < 0.9: good reliability, 0.7 < 0.8: acceptable reliability, 0.6 < 0.7: questionable reliability, 0.5 < 0.6: poor reliability, < 0.5: unacceptable reliability, 0: no reliability. On this scale, a correlation of .9(90%) would indicate a very high correlation (good reliability) and a value of 10% a very low one (poor reliability).

CONTACTS AND LOCATIONS:
Overall Officials: Nukusbekova, Principal Investigator — Doctor
Locations (2):
- Kazakhstan (2):
  - SOS Medical Assistance, Almaty
  - V-ent, Almaty

IPD SHARING:
Plan to Share IPD: Yes
Non-identifiable IPD will be shared upon request with all required information
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be available upon completion of the study primary analysis
Access Criteria: Only people with access will be able to see the data